CLINICAL TRIAL: NCT00834743
Title: A Two-Way Crossover, Open-Label, Single-Dose, Fasting, Bioequivalence Study of Metformin ER 750 mg Tablets Versus Glucophage® XR 750 mg Tablets in Normal Healthy Non-smoking Male and Female Subjects
Brief Title: Metformin ER 750 mg Tablets, Fasting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2734
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Metformin ER 750 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: Glucophage® XR 750 mg Tablets

INTERVENTIONS:
Drug: Glucophage® XR 750 mg Tablets — 1 x 750 mg, single-dose fasting
  Arms: 2
Drug: Metformin ER 750 mg Tablets — 1 x 750 mg, single-dose fasting
  Arms: 1

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of metformin from a test formulation of Metformin ER 750 mg Tablets versus the reference Glucophage® XR 750 mg Tablets under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female with a minimum age of 18 years (i.e. non-smoker or non-tobacco user for at least 90 days prior to pre-study medical screening).
* Body Mass Index (BMI - weight/height²) greater than or equal to 19 kg/m² and less than or equal to 30 kg/m².
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.
* Normal findings in the physical examination, 12-lead ECG and vital signs (blood pressure between 100-140/60-90 mmHg, heart rate between 50-99 beats/min, temperature between 35.8ºC and 37.5ºC).
* Negative for drugs of abuse, nicotine, alcohol, hepatitis B-surface antigen, hepatitis C and HIV, and for female subjects, pregnancy (serum ß-CG).
* No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides they are not clinically significant.
* Female subjects who are surgically sterile for at least six months or post-menopausal for at least one year, or who will avoid pregnancy prior to the study, during the study and up until one month after the end of the study.

Exclusion Criteria:

* Known history of hypersensitivity to metformin (e.g. Glucophage®) and/or related drugs such as glyburide (Diaβeta®, Euglucon®), tolbutamide (Orinase®, Apo-chlorpropamide), acetohexamide (Dimelor®), chlorpropamide (Diabinese®) and glipizide (Glucotrol®, Glibenese®).
* Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurologic, hematological, liver, or kidney disease unless judged no clinically significant by the Principal Investigator, or medical designate.
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness during the last four weeks prior to entry into this study.
* Presence of any significant physical or organ abnormality.
* Any subject with a history of drug abuse.
* Any psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator, or medical designate.
* Use of any prescription medication within 14 days preceding entry into this study.
* Use of over-the-counter (OTC) medication within seven days preceding entry into this study (except for spermicidal/barrier contraceptive products).
* Female subjects: use of oral contraceptives or contraceptive implants (Such as Norplant®) within 30 days prior to drug administration or a depot injection of progestogen drug (e.g. Depro-Provera®) within one year prior to drug administration.
* Female subjects: presence of pregnancy or lactation.
* Any subject who has had blood withdrawn within 56 days preceding this study, taken during the conduct of any clinical study at a facility other than BCR, or within the lockout period specified by a previous study conducted at BCR.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* Any subject who has donated blood within 56 days preceding this study.
* Any subject who has participated as a plasma donor in a plasmapheresis program within seven days preceding this study.
* Significant or recent history of asthma (After 12 years of age).
* Any subject with a recent (less than one year) history of alcohol abuse.
* Intolerance to venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-08; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y. Tam, M.D., Principal Investigator — Biovail Contract Research
Locations (1):
- Biovail Contract Research, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Metformin) First: 750 mg Metformin Extended Release Tablets test product dosed in first period followed by 750 mg Glucophage® XR Tablets reference product dosed in the second period.
- Reference (Glucophage®) First: 750 mg Glucophage® XR Tablets reference product dosed in first period followed by 750 mg Metformin Extended Release Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Metformin) First | Reference (Glucophage®) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Test (Metformin) First | Reference (Glucophage®) First
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test (Metformin) First | Reference (Glucophage®) First
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Metformin) First | Reference (Glucophage®) First | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 2
  Black | 2 | 4 | 6
  White | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Metformin): 750 mg Metformin Extended Release Tablets test product dosed in either period.
- Reference (Glucophage®): 750 mg Glucophage® XR Tablets reference product dosed in either period.
Arm/Group | Test (Metformin) | Reference (Glucophage®)
Number analyzed (Participants) | 31 | 31
ng/mL | 875.86 (276.2) | 886.39 (297.74)
Statistical Analysis 1: Comparison: Test (Metformin) vs Reference (Glucophage®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 99.49, 90% CI [90.65 to 109.18] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Metformin) | Reference (Glucophage®)
Number analyzed (Participants) | 31 | 31
ng*h/mL | 6068.12 (2052.11) | 6188.74 (2293.91)
Statistical Analysis 1: Comparison: Test (Metformin) vs Reference (Glucophage®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99, 90% CI [91.44 to 107.19] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 36 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Metformin) | Reference (Glucophage®)
Number analyzed (Participants) | 31 | 31
pg*h/mL | 6301.73 (2175.6) | 6495.16 (2442.93)
Statistical Analysis 1: Comparison: Test (Metformin) vs Reference (Glucophage®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 99.05, 90% CI [90.57 to 108.32] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.